CLINICAL TRIAL: NCT06792812
Title: The Impact of Ginger Mouthwash on the Pregnant Women With Stress and Gingivitis by Measuring Different Salivary Biomarkers Levels (Randomized Clinical Trial)
Brief Title: The Impact of Ginger Mouthwash on the Pregnant Women With Stress and Gingivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Batool Abbas Tareq, Principal Investigator, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MUOSU-202125
Record Dates: First submitted 2024-10-09; First posted 2025-01-27 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Mouth Diseases; Bleeding Gum; Stress
Keywords: gingivitis; stress; pregnancy; ginger mouthwash
MeSH Terms: conditions — Mouth Diseases; Gingival Hemorrhage; Gingivitis

STUDY DESIGN:
Intervention Model Description: pregnant with stress and gingivitis, will be selected and enrolled in this study. Subsequently, subjects will be equally divided and randomly allocated into three groups, each group receiving a similar number of subjects (n=18)
Who Masked: Participant, Care Provider, Investigator
Masking Description: the products will be packaged in such a way that they are not recognizable by the operator or the patient. Each package will be assigned a number that in turn will refer to the type of the product. The association between the number and type of the product will be collected by another operator according to the association carried out by a dedicated software. The operator who will deliver the product will be informed about the type only at the end of the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ginger mouthwash (Experimental): Ginger mouthwash (Pasta del Capitano) Participants will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. participants will be received a toothbrush with medium-hardness bristles and a toothpaste (COLGATE) and all participants are instructed to decrease stress by a combination of diaphragmatic breathing and muscle relaxation. No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 7 days.
  Interventions: Drug: ginger mouthwash
- chlorohexidine mouthwash (Experimental): Chlorhexidine 0.12% Participants will be given as positive control the Chlorhexidine 0.12%, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. participants will be received a toothbrush with medium-hardness bristles and a toothpaste (COLGATE) and all participants are instructed to decrease stress by a combination of diaphragmatic breathing and muscle relaxation. No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 7 days.
  Interventions: Drug: chlorohexidine mouthwash
- placepo (Experimental): Placebo Product Participants will be given distilled water, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. participants will be received a toothbrush with medium-hardness bristles and a toothpaste (COLGATE)and all participants are instructed to decrease stress by a combination of diaphragmatic breathing and muscle relaxation. No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ginger mouthwash — contain Sulfetal Zn® (Zinc Coco Sulphate) has a cleansing and antibacterial action and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. participants will be received a toothbrush with medium-hardness bristles and a toothpaste (COLGATE)and all participants are instructed to decrease stress by a combination of diaphragmatic breathing and muscle relaxation. No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 7 days.
  Arms: ginger mouthwash
Drug: chlorohexidine mouthwash — Subjects will then be given Chlorhexidine 0.12%mouthwash, as an active comparator, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. participants will be received a toothbrush with medium-hardness bristles and a toothpaste (COLGATE)and all participants are instructed to decrease stress by a combination of diaphragmatic breathing and muscle relaxation. No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 7 days.
  Arms: chlorohexidine mouthwash
Drug: Placebo — Subjects will be given the nonactive control, distilled water, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. participants will be received a toothbrush with medium-hardness bristles and a toothpaste (COLGATE)and all participants are instructed to decrease stress by a combination of diaphragmatic breathing and muscle relaxation. No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 7 days.
  Arms: placepo

SUMMARY:
The study aims to determine ginger mouthwash's impact on gingival health, IL-6, cortisol, LF, and 8-OHdG levels in pregnant women with stress and gingivitis compared to CHX and distilled water.

Objectives:

1. Evaluate the clinical efficiency of ginger mouth rinse for 7 days to control gingival inflammation by measuring the clinical periodontal parameters, Plaque Index (PI), Gingival Index (GI), and Bleeding on probing (BOP) in comparison with CHX and placebo mouth rinses in pregnant women who have stress and gingivitis.
2. Measuring salivary IL_6, Cortisol, LF, and 8-OHdG levels by Enzyme-linked immunosorbent assay (ELISA) at the baseline visit before and after 7 days of using ginger mouth rinse compared to CHX and placebo mouth rinses.
3. Assessment of participants' feedback regarding ginger, CHX, and placebo mouth rinses after 7 days of use by Visual Analog Scale (VAS) questionnaire.
4. correlate IL_6, Cortisol, LF and 8-OHdG salivary levels with clinical periodontal parameters (GI, BOP, PI) to assess their relationship in pregnant women with stress and gingivitis.

DETAILED DESCRIPTION:
54 pregnant with stress will be enrolled, who show with gingivitis The investigator assesses symptoms of stress using a translated Arabic version of Perceived Stress Scale (PSS) Each pregnant answers following questions Questions never almost never sometimes fairly often very often

1. In the last month how often have you been upset because of something that happened unexpectedly?
2. In the last month, how often have you felt that you were unable to control the important things in your life
3. In the last month, how often have you felt nervous and stressed?
4. In the last month, how often have you felt confident about your ability to handle your personal problems?
5. In the last month, how often have you felt that things were going your way?
6. In the last month, how often have you found that you could not cope with all the things that you had to do?
7. In the last month, how often have you been able to control irritations in your life?
8. In the last month, how often have you felt that you were on top of things
9. In the last month, how often have you been angered because of things that happened that were outside of your control?
10. In the last month, how often have you felt difficulties were piling up so high that you could not overcome them?

For each question choose from the following alternatives:

0 - never 1 - almost never 2 - sometimes 3 - fairly often 4 - very often Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.

* Scores ranging from 0-13 would be considered low stress.
* Scores ranging from 14-26 would be considered moderate stress.
* Scores ranging from 27-40 would be considered high perceived stress.

A triple-blind, randomized parallel 3-arms clinical trial include using the following mouth rinses, 0.12% CHX (KIN Gingival, KIN, Barcelona, Spain) as positive-control, distilled water (placebo, nonactive control) with food additives (to blind the subjects and examiner) and ginger mouthwash (Pasta del Capitano, Italy)

The examiner will perform randomization for the enrollment patients in 3 groups. Each group will be assigned a letter (A, B, or C) corresponding to the intervention used. Random numbers were generated and used to re-sort the order of the groups and participants (n=54), who will be distributed into designated groups, each group received a similar number of subjects (n=18) , by using a Microsoft Excel random table (Microsoft Office 2021, Microsoft Corporation, USA). Then, coded bottles with the interventions will be delivered to the participants together with instructions for use.

The participants will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. Discontinuation of the mouthwash will be advised in cases of any allergic reaction. All participants will be received a toothbrush with medium-hardness bristles and a toothpaste, and All participants are instructed to decrease stress by a combination of diaphragmatic breathing and muscle relaxation Saliva collection for IL-6, cortisol, lactoferrin, and 8-OHdG measurement then clinical periodontal parameters examination starting with gingival index designed to assess the severity and quality of gingival inflammation in an individual or population. The gingival inflammation is assessed on the basis of color, consistency and bleeding on probing. A periodontal probe will be runned along the gingival margin. The gingiva surrounding the tooth is assessed at four sites: mesio-facial papilla, facial marginal gingiva, disto-facial papilla and lingual marginal gingiva.

Followed by dryness and wait then measurement of BOP for the six surfaces of all teeth except wisdom teeth through gently inserting the periodontal probe to the depth of the gingival sulcus then removed coronally and waited for 30 s to observe the presence of bleeding (0=no bleeding, 1=presence of bleeding)

Then finally followed by the Plaque Index :

A periodontal probe may be used to confirm the presence of plaque. Scores were recorded on four surfaces; distal, mid, and mesial points on the facial (buccal) and lingual (palatal) aspects. as follows:

0- ne plaque (left blank)

1- plaque present ( recorded)

First visit after 7 days, from the baseline visit. Saliva collection and clinical periodontal parameters scoring (GI, BOP, PI) will be performed again as described at baseline visit. The mouthwash bottles will be retrieved, and the remaining volume will be determining to further evaluate the compliance with mouth rinsing. For the purpose of self-assessment, a visual analog scale (VAS)- score based questionnaire was filled out by each participant at the end of the trial to evaluate the intervention. The questionnaire and method of data interpretation were adopted and modified from a previous study

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant with gingivitis with impact periodontium.
2. Pregnant with stress.
3. Pregnant in 5,6,7 months.
4. Pregnant in age (20-30) years old.
5. Good general health without systemic disease.
6. The presence of at least 20 or more natural teeth.
7. No antibiotic therapy has been received in the last 3 months.

Exclusion Criteria:

1. currently use any mouthwash.
2. Pregnant who rejects the form of informed approval.
3. Pregnant with dental implants and orthodontic or prosthodontic appliances or any retentive factor of dental plaque.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 0-7 days
  Measuring Change in the clinical periodontal parameter (Bleeding on Probing) Subjects will undergo the measurement bleeding on probing for the six surfaces of all teeth except wisdom teeth through gently inserting the periodontal probe to the depth of the gingival sulcus then removed coronally and waited for 30 s to observe the presence of bleeding (0=no bleeding, 1=presence of bleeding).

SECONDARY OUTCOMES:
Secondary Outcome Measure | 0-7 days
  Measurement changes in salivary Interleukin 6 by using Enzyme-linked immunosorbent assay (ELISA) before and after using mouthwash by saliva collection before and after using mouthwash Sensitivity 0.94 pg/mL Detection Range 1.56-100 pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Batool Alshuwaili, B.D.S, Principal Investigator — Al-Mustansiriyah University
Locations (1):
- Mustansiriyah University, Baghdad, Iraq